CLINICAL TRIAL: NCT06011447
Title: The Use of Laser Speckle Imaging in the Evaluation of Successful Revascularisation of Patients With Ischemic Tissue Loss
Brief Title: Laser Speckle Imaging in Ischaemic Tissue Loss
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: VS20/130302
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetes and wound ulcers
  Interventions: Other: Device to view the skin

INTERVENTIONS:
Other: Device to view the skin — Application of device to help view the wound area better

SUMMARY:
Peripheral arterial disease is a condition in which the arteries become narrowed due to a build up of cholesterol, as a result, blood cannot flow efficiently through the arteries and this can compromise the parts of the body supplied by these arteries. In its most severe form, peripheral arterial disease can lead to decomposition of tissues in the feet, leading to ulcers or gangrene. Patients with peripheral arterial disease undergo procedures to improve blood flow.

However, there are often multiple arteries to treat and each intervention carries risk. It therefore can be difficult to judge how much treatment is sufficient to promote healing. Laser Speckle Imaging is a technique used to demonstrate blood flow in the skin. It is hoped that changes in skin blood flow, as measured by LSI, immediately after a procedure to improve blood flow, may help in the decision making as to whether further intervention is necessary. An LSI scan will be performed before a procedure for tissue loss and immediately after it is performed. The patient's clinical records will then be checked to see whether the wound has improved and whether the difference in LSI scans correlated with this.

ELIGIBILITY:
Inclusion Criteria:

Patients with diabetes Patients with a foot ulcer or open wound Patients aged over 18 Patients able to given consent Patients undergoing femoropopliteal bypass or superficial femoral / popliteal artery angioplasty

Exclusion Criteria:

nability to consent Planned major limb amputation for the affected limb

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with vascular ulcers
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
fail to heal wounds | 7 months
  The study aims to assess whether wounds which fail to heal are associated with small differences in LSI blood flow measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds NHS Teaching Hospitals, Leeds, United Kingdom